CLINICAL TRIAL: NCT03878576
Title: The Effect of Content of Barley Beta-glucans in Bread on Postprandial Blood Sugar
Acronym: ARRS-bGL-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Community Health Centre Ljubljana (Other); Slovenian Research Agency (Other); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KME/0120-441/2018/4
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Glycemic Index
Keywords: Glycemic Index; glycemic response; bread; barley; beta-glucans; glucose level; continous glucose monitoring
MeSH Terms: interventions — I-kappa B Kinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- REFERENCE: white bread - BGL0 [RP] (Active Comparator): Participants consume a meal of bread BGL0 standardised to contain 25 g of available carbohydrates. Sample consumed together with 300 mL of water in up to 15 minutes.
  Interventions: Other: REFERENCE: white bread - BGL0 [RP]
- TEST: b-glucan enriched bread - BGL2 [IP1] (Experimental): Participants consume a meal of bread BGL2 standardised to contain 25 g of available carbohydrates. Sample consumed together with 300 mL of water in up to 15 minutes.
  Interventions: Other: TEST: b-glucan enriched bread - BGL2 [IP1]
- TEST: b-glucan enriched bread - BGL3 [IP2] (Experimental): Participants consume a meal of bread BGL3 standardised to contain 25 g of available carbohydrates. Sample consumed together with 300 mL of water in up to 15 minutes.
  Interventions: Other: TEST: b-glucan enriched bread - BGL3 [IP2]
- TEST: b-glucan enriched bread - BGL4 [IP3] (Experimental): Participants consume a meal of bread BGL4 standardised to contain 25 g of available carbohydrates. Sample consumed together with 300 mL of water in up to 15 minutes.
  Interventions: Other: TEST: b-glucan enriched bread - BGL4 [IP3]

INTERVENTIONS:
Other: REFERENCE: white bread - BGL0 [RP] — Determination of glycemic response after consumption of BGL0.
  Arms: REFERENCE: white bread - BGL0 [RP]
Other: TEST: b-glucan enriched bread - BGL2 [IP1] — Determination of glycemic response after consumption of BGL0.
  Arms: TEST: b-glucan enriched bread - BGL2 [IP1]
Other: TEST: b-glucan enriched bread - BGL3 [IP2] — Determination of glycemic response after consumption of BGL0.
  Arms: TEST: b-glucan enriched bread - BGL3 [IP2]
Other: TEST: b-glucan enriched bread - BGL4 [IP3] — Determination of glycemic response after consumption of BGL0.
  Arms: TEST: b-glucan enriched bread - BGL4 [IP3]

SUMMARY:
The effect of content of barley beta-glucans in bread on postprandial blood sugar will be measured with open-label crossover study. Study will be conducted in Slovenia on 10-12 adult subjects who will test three barley beta-glucan containing bread formulations (food) in comparison with a reference white bread. Objective of the study is to investigate the influence of the content of barley beta-glucan in bread on glycaemic index (incremental area under the curve (IAUC) for the blood glucose response curve for barley beta-glucan containing breads in comparison to reference white bread.

ELIGIBILITY:
Inclusion Criteria:

* Subject Informed consent form (ICF) is singed
* Aged above 18 years at the time of the signature of ICF
* No known food allergy or intolerance
* No medications known to affect glucose tolerance - stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable.
* Willing to follow all study procedures, including attending all site visits (including sessions for blood sampling and use of CGM)
* Body mass index (BMI) > 25

Exclusion Criteria:

* Subject Informed consent form (ICF) is singed
* Aged above 18 years at the time of the signature of ICF
* No known food allergy or intolerance
* No medications known to affect glucose tolerance - stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable.
* Willing to follow all study procedures, including attending all site visits (including sessions for blood sampling and use of CGM)
* Body mass index (BMI) > 25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Change in glycaemic response (capillary blood glucose) | 2 hours
  Change in incremental area under the curve (IAUC) the blood glucose response curve for barley beta-glucan containing breads (investigational products; IP1-3), in comparison to white bread (reference product; RP)

OTHER OUTCOMES:
Glucose level as measured with continuous glucose monitor (CGM) | up to 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, PhD, Study Chair — Institut za nutricionistiko
Locations (1):
- Nutrition Institite, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No